CLINICAL TRIAL: NCT04630795
Title: An Investigation Into the Efficacy of a Patient-specific Turf-Like Insole in Reducing Plantar Pressure and Improving Skin Microcirculation in Patients With Diabetic Neuropathy.
Brief Title: ViscoTurf - Preventing Secondary Diabetic Foot Ulceration.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Staffordshire University (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Roozbeh Naemi, Professor in Biomechanics, Staffordshire University
Other Study IDs: SU-20-001
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Foot
Keywords: Biomechanics, perfusion, plantar soft tissue, skin microcirculation,
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3D printed insole: Intervention insole will be produced as 3D printed insole with the Turf-Like patches incorporated in the areas of interest, while the Control Insole will be a standard 3D printed flat insole with NO Turf-like patches.
  Interventions: Device: ViscoTurf insole; Device: Control insole

INTERVENTIONS:
Device: ViscoTurf insole — Intervention insole will be produced as 3D printed insole with the Turf-Like patches incorporated in the areas of interest.
  Other Names: Turf like insole
Device: Control insole — Control Insole will be a standard 3D printed flat insole with NO Turf-like patches.
  Other Names: Standard insole

SUMMARY:
Diabetic Foot Ulceration (DFU) is one of the most common complication of diabetes costing the NHS over £970m annually. Management of foot ulcers is time-consuming and expensive with 45% taking more than six months to heal. Around 25% of patients re-ulcerate in 3 months, 40% within 1 year and 60% within 3 years and patients who have achieved wound closure are generally considered to be in remission rather than healed. A patient presenting with a foot ulcer has a greatly elevated risk of amputation while 80% of amputations can be prevented with the appropriate treatment, such as footwear intervention.

ViscoTurf is a novel, 3D printed, orthotic device designed specifically for this purpose. It emulates the function of natural turf to provide cushioning, optimised offloading and better microcirculation on the vulnerable areas of the plantar surface of the foot. This improves perfusion (the delivery of blood to the capillary bed) in the load bearing regions of the foot where the risk of re-ulceration is very high. An earlier feasibility study established proof-of-concept, showing ViscoTurf achieved a higher and longer-lasting increase in perfusion compared to conventional support structures. ViscoTurf insoles can be automatically designed to the foot size and 3D printed.

The main purpose of this study is to investigate the immediate effect of walking in Viscoturf insole (Turf-Like insoles) on skin perfusion and pressure at the sole of the foot in diabetic patients with history of ulceration. To achieve this, the immediate efficacy (effect as a result of walking for 15 meters) of Viscoturf insole will be assessed and compared to that of the standard flat insole. Intervention insole will be produced as 3D printed insole with the Turf-Like patches incorporated in the areas of interest, while the Standard Insole will be a standard 3D printed flat with NO Turf-like patches.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 OR Type 2 diabetes
* Over 18
* History of foot ulcer

Exclusion Criteria:

* History of recent major lower limb surgery (amputation) or revascularisation and orthopaedic reconstruction over the last 3 months
* Current active foot ulcer
* Not be able to walk unassisted for 15 meters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are selected from patients of King's diabetic foot clinic who meet the inclusion/exclusion criteria and who are consent to take part.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Plantar skin perfusion before and after use. | March-July 2021
  The primary outcome measure is the improvement in plantar skin perfusion, which is the difference between skin perfusion before and after use.

SECONDARY OUTCOMES:
Plantar Pressure during walking | March-July2021
  The secondary outcome measure is plantar pressure underneath the critical areas when walking in the insole.

IPD SHARING:
Plan to Share IPD: No
Participants with diabetes will be recruited from Kings College Hospital Trust (KCHT) using the inclusion and exclusion criteria previously outlined. A dedicated research podiatric practitioner nurse will first identify the patients who meet the inclusion exclusion criteria by searching through the KCHT diabetic foot patient database and clinical records.